CLINICAL TRIAL: NCT02716987
Title: A Phase 1, Open-Label, Positron Emission Tomography Study in Healthy Subjects to Determine D-Amino Acid Oxidase Brain Enzyme Occupancy of TAK-831 After Single-Dose Oral Administration in Healthy Subjects
Brief Title: Study to Determine D-amino Acid Oxidase Brain Enzyme Occupancy of TAK-831 After Single-dose Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-831-1003; 2015-004509-17 (EudraCT Number); U1111-1176-7493 (Registry Identifier: WHO); 15/LO/1916 (Registry Identifier: NRES)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Set A: TAK-831 100 mg (Experimental): TAK-831 100 milligram (mg), suspension, orally, once on Day 1 and up to 100 megabecquerel (MBq) of Positron Emission Tomography (PET) ligand PGM028299 labeled with [18F] ([18F]PGM299) with a maximal mass up to 12.5 microgram (mcg), injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
  Interventions: Drug: TAK-831; Drug: [18F]PGM299
- Set A: TAK-831 200 mg (Experimental): TAK-831 200 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
  Interventions: Drug: TAK-831; Drug: [18F]PGM299
- Set A: TAK-831 250 mg (Experimental): TAK-831 250 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
  Interventions: Drug: TAK-831; Drug: [18F]PGM299
- Set A: TAK-831 500 mg (Experimental): TAK-831 500 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
  Interventions: Drug: TAK-831; Drug: [18F]PGM299
- Set B: [18F]PGM299 (Experimental): [18F]PGM299 up to 100 MBq (with a maximal mass up to 12.5 mcg), injection, intravenously, prior to PET imaging on Days 1 and 10.
  Interventions: Drug: [18F]PGM299

INTERVENTIONS:
Drug: TAK-831 — TAK-831 oral suspension.
  Arms: Set A: TAK-831 100 mg; Set A: TAK-831 200 mg; Set A: TAK-831 250 mg; Set A: TAK-831 500 mg
Drug: [18F]PGM299 — [18F]PGM299 injection

SUMMARY:
The purpose of this study is to determine the relationship between TAK-831 dose, plasma exposure, extent and duration of brain D-amino acid oxidase (DAO) enzyme occupancy following single oral dosing of TAK-831 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831. TAK-831 is a highly selective and potent inhibitor of DAO, a peroxisomal enzyme active towards neutral D-amino acids which potentially effects cerebellar dysfunction. This study will look at the relationship between TAK-831 plasma exposure and the extent and duration of brain DAO enzyme occupancy after single oral dosing of TAK-831 in healthy male participants using [18F]PGM299 radioactive tracer injection and PET imaging.

The study will enroll up to 22 participants in two different sets. Up to 16 participants will be enrolled in Set A. Within that total, up to 5 dose levels of TAK-831 may be evaluated, with up to 6 participants per dose level, although typically, there will be 2 to 3 participants per dose level. All participants in Set A will also receive up to 3 doses of [18F]PGM299. Up to 6 participants will be enrolled in Set B. All participants in Set B will be assigned to single treatment group to receive 2 doses of [18F]PGM299.

All participants in Set A will be asked to take single oral dose of TAK-831 suspension on Day 1. In Set A, each of the participant will receive a maximum of 3 PET scans with [18F]PGM299; 1 at baseline 2 following a single oral dose of TAK-831 on Days 1 and 2. In Set B, each of the participant will receive 2 PET scans with [18F]PGM299 on Days 1 and 10. Set B will be conducted after the confirmation of blockade of [18F]PGM299 binding by TAK-831 in 2 to 4 participants of Set A.

This multi-center trial will be conducted in the United Kingdom. The overall time to participate in this study is 62 days. Participants in Set A will make 4 visits to the clinic, and participants in Set B will make 3 visits to the clinic and all will be contacted by telephone on Day 15 (Set A) and Day 12 (Set B) of treatment period for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is in good health as determined by physical examination, electrocardiogram (ECG), and laboratory evaluations.
4. Is a healthy male aged 25 to 55 years, inclusive, at the time of informed consent and first injection of the PET tracer.
5. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive, at Screening.
6. Agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose.

Exclusion Criteria:

1. Has received any investigational compound or device within 3 months or 5 half-lives, whichever is longer, prior to Check-in for Screening.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant (CS), neurologic (including seizure disorder), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal (GI), urologic, immunologic, or endocrine disease or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. Has a known hypersensitivity to any component of the formulation of TAK-831 or related compounds, or to [18 F]PGM299 or to any of its components.
5. Has a positive urine or breath test result for drugs of abuse (defined as any illicit drug use), ethanol (alcohol), or cotinine at Screening, Check-in for Baseline Imaging/Confinement Period 1, or Check-in for the Treatment/Confinement Period 2 (Day -1) for a participant participating in Set A or at Screening, Check-in for Tracer TEST PET Imaging/Confinement Period 1, or Check-in for RE-TEST PET Imaging/Confinement Period 2 for a participant participating in Set B.
6. Has a history of drug abuse (defined as any illicit drug use) or a history of ethanol (alcohol) abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from ethanol (alcohol) and drugs throughout the study.
7. Has taken any medication, supplements, or food products during the time periods listed in the excluded medications and dietary products table.
8. Intends to donate sperm during the course of this study or for 90 days after the last dose of study medication.
9. Has evidence of current cardiovascular, central nervous system, hepatic, or hematopoietic disease; renal, metabolic or endocrine dysfunction; serious allergy, asthma, hypoxemia, hypertension, or allergic skin rash; or there is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-831 or a similar drug in the same class, which might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease and cardiac arrhythmias.
10. Has current or recent (within 6 months) GI disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption), any surgical intervention known to impact absorption (example, bariatric surgery or bowel resection), esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent (more than once per week) occurrence of heartburn.
11. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
12. Has a positive test result for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody (HCAB), or human immunodeficiency virus (HIV) infection at Screening.
13. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 44 days prior to Check-in for Confinement Period 1. Cotinine test is positive at Screening, or Check-in for Confinement Period 1, or Confinement Period 2.
14. Has poor peripheral venous access.
15. Has an abnormal Allen's test in either upper extremity.
16. Has donated or lost 450 milliliter (mL) or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Confinement Period 1.
17. Has an abnormal CS ECG at Screening, Check-in for Confinement Period 1, or at Check-in for Confinement Period 2. Entry of any participant with an abnormal (not clinically significant [NCS]) ECG must be approved and documented by signature of the coordinating investigator or delegate.
18. Has a supine blood pressure outside the ranges of 100 to 140 millimeter of mercury (mm Hg) for systolic and 50 to 90 mm Hg for diastolic, confirmed with 1 repeat testing within a maximum of 30 minutes, at the Screening Visit, Check-in for Confinement Period 1, or Confinement Period 2.
19. Has a resting heart rate outside the range of 50 to 90 beats/minute, confirmed with 1 repeat testing within a maximum of 30 minutes, at the Screening Visit, Check-in for Confinement Period 1, or Confinement Period 2.
20. Has a Fridericia's Correction Formula (QTcF) - QTcF interval greater than (>) 450 millisecond (msec) or PR outside the range of 120 to 220 msec, confirmed with 1 repeat testing within a maximum of 30 minutes, at the Screening Visit, Check-in for Confinement Period 1, or Confinement Period 2.
21. Has abnormal Screening laboratory values that suggest a CS underlying disease or the following laboratory abnormalities: Alanine Aminotransferase (ALT) and/or Alanine serum transaminase AST >1.5*upper limit of normal (ULN).
22. Has a risk of suicide according to the investigator's clinical judgment (example, per Columbia-Suicide Severity Rating Scale [C-SSRS]) or has made an attempt in the previous 6 months.
23. Has had a seizure or convulsion (lifetime), including absence seizure and febrile convulsion.
24. In the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.
25. Has had previous exposure to ionizing radiation such that, in combination with the exposure from this study, their exposure will be >10 millisievert (mSv) for the previous year.
26. Has a contraindication to medical resonance imaging (MRI) based on the standard MRI screening questionnaire. Contraindications include ferromagnetic foreign bodies (example, shrapnel, ferromagnetic fragments in the orbital area), certain implanted medical devices (example, aneurysm clips, cardiac pacemakers) or claustrophobia.
27. Has findings on screening brain MRI scan that will potentially compromise participant safety or the scientific integrity of the study data, if the participant were to participate in this study.
28. Has prolonged prothrombin time (PT) or activated partial thromboplastin time (PTT) or reduced platelet count (less than [<] 100*10^9/Liter [L]).

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United Kingdom from 21-Mar-2016 to 30-Aug-2016.
Pre-assignment Details: Healthy participants in Set A received up to 100 megabecquerel (MBq) of [18F]PGM299 for 3 PET scans at baseline, 2, and 26 hours post TAK-831. Set A participants also received a single dose of TAK-831 (100 milligram [mg], 200 mg, 250 mg, or 500 mg). Healthy participants in Set B received up 100 MBq of [18F]PGM299 for 2 PET scans on Day 1 and 10.
Groups:
- Set A: TAK-831 100 mg: TAK-831 100 mg, suspension, orally, once on Day 1 and up to 100 MBq of Positron Emission Tomography (PET) ligand PGM028299 labeled with [18F] ([18F]PGM299) with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
- Set A: [18F]PGM299 Baseline: [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline only. Participant in this reporting group discontinued from the study and did not receive any TAK-831 dose.
Period: Overall Study
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg | Set B: [18F]PGM299 | Set A: [18F]PGM299 Baseline
Started | 4 | 2 | 5 | 2 | 6 | 1
Completed | 4 | 2 | 4 | 2 | 5 | 0
Not Completed | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Ligand synthesis failure | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled and received an investigational drug ([18F]PGM299 or TAK-831).
Groups:
- Set A: TAK-831 100 mg: TAK-831 100 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
- Total: Total of all reporting groups
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg | Set B: [18F]PGM299 | Set A: [18F]PGM299 Baseline | Total
Number analyzed (Participants) | 4 | 2 | 5 | 2 | 6 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 5 | 2 | 6 | 1 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 2 | 5 | 2 | 6 | 1 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 4 | 0 | 6
  White | 3 | 2 | 3 | 1 | 2 | 1 | 12
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 4 | 2 | 5 | 2 | 6 | 1 | 20
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 4 | 2 | 3 | 2 | 4 | 1 | 16
  Ex-smoker | 0 | 0 | 2 | 0 | 2 | 0 | 4
Alcohol Classification [Count of Participants; unit: Participants]
  Never drunk | 0 | 0 | 2 | 1 | 1 | 1 | 5
  Current drinker | 3 | 2 | 3 | 1 | 3 | 0 | 12
  Ex-drinker | 1 | 0 | 0 | 0 | 2 | 0 | 3
Caffeine Consumption [Count of Participants; unit: Participants]
  Caffeine consumption | 4 | 2 | 5 | 2 | 3 | 1 | 17
  No caffeine consumption | 0 | 0 | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Distribution (VT) of [18F]PGM299 in the Cerebellar Grey Matter (GM) for Each PET Scan
Time Frame: Set A: Baseline (PET scan 1), 2 hours (PET scan 2) and 26 hours (PET scan 3) post-TAK-831 dose; Set B: Day 1 (PET scan 1) and Day 10 (PET scan 2)
Population: The set included all participants who had at least 1 technically adequate PET scan.
Measure: Number; unit: milliliter per cubic centimeter(mL/cm^3)
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg | Set B: [18F]PGM299 | Set A: [18F]PGM299 Baseline
Number analyzed (Participants) | 4 | 2 | 5 | 2 | 6 | 1
milliliter per cubic centimeter(mL/cm^3)
  Participant 1- PET Scan 1 | 1.211 | 1.247 | 1.349 | 1.683 | 0.658 | 0.863
  Participant 1- PET Scan 2 | 0.400 | 0.126 | 0.247 | 0.114 | 1.109 | NA — Data not reported because participant discontinued the study after Baseline PET scan 1.
  Participant 1- PET Scan 3 | 1.467 | 0.543 | 0.58 | 1.182 | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data not reported because participant discontinued the study after Baseline PET scan 1.
  Participant 2- PET Scan 1 | 0.663 | 1.585 | 0.743 | 2.095 | 0.884 | NA — Data was not reported because only one participant was included in this arm.
  Participant 2- PET Scan 2 | 0.241 | 0.217 | 0.266 | 0.172 | 1.130 | NA — Data was not reported because only one participant was included in this arm.
  Participant 2- PET Scan 3 | 0.809 | 0.77 | 0.425 | 0.553 | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 3- PET Scan 1 | 1.397 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.981 | NA — Data was not reported because only two participants were enrolled in this arm. | 1.504 | NA — Data was not reported because only one participant was included in this arm.
  Participant 3- PET Scan 2 | 0.858 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.189 | NA — Data was not reported because only two participants were enrolled in this arm. | 1.388 | NA — Data was not reported because only one participant was included in this arm.
  Participant 3-PET Scan 3 | 1.078 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.802 | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 4- PET Scan 1 | 1.297 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.853 | NA — Data was not reported because only two participants were enrolled in this arm. | 1.459 | NA — Data was not reported because only one participant was included in this arm.
  Participant 4- PET Scan 2 | 0.592 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.254 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.979 | NA — Data was not reported because only one participant was included in this arm.
  Participant 4-PET Scan 3 | 1.055 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.67 | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 1 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 0.976 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.895 | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 2 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — PET scan 2 was not performed due to ligand synthesis failure. | NA — Data was not reported because only two participants were enrolled in this arm. | 1.077 | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 3 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — PET scan 3 was not performed due to ligand synthesis failure. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 6- PET Scan 1 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only five participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 1.036 | NA — Data was not reported because only one participant was included in this arm.
  Participant 6 -PET Scan 2 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only five participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data is not available because this participant withdrew the study after PET Scan 1. | NA — Data was not reported because only one participant was included in this arm.

2. Primary Outcome: Non-displaceable Binding Potential (BPND) of [18F]PGM299 in the Cerebellar GM for Each PET Scan
Time Frame: as for outcome 1
Population: The set included all participants who had at least 1 technically adequate PET scan.
Measure: Number; unit: ratio
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg | Set B: [18F]PGM299 | Set A: [18F]PGM299 Baseline
Number analyzed (Participants) | 4 | 2 | 5 | 2 | 6 | 1
ratio
  Participant 1- PET Scan 1 | 10.99 | 7.31 | 6.71 | 8.96 | 3.77 | 5.49
  Participant 1- PET Scan 2 | 3.26 | -0.28 | 0.47 | -0.20 | 4.99 | NA — Data not reported because participant discontinued the study after Baseline PET scan 1.
  Participant 1- PET Scan 3 | 7.89 | 4.22 | 4.32 | 11.19 | NA — Data not reported since only PET Scan 1 and 2 were planned to be analysed in Set B. | NA — Data not reported because participant discontinued the study after Baseline PET scan 1.
  Participant 2- PET Scan 1 | 3.88 | 8.38 | 3.53 | 13.35 | 13.49 | NA — Data was not reported because only one participant was included in this arm.
  Participant 2- PET Scan 2 | 1.01 | 0.16 | 0.25 | 0.06 | 5.89 | NA — Data was not reported because only one participant was included in this arm.
  Participant 2- PET Scan 3 | 4.39 | 6.06 | 2.17 | 4.59 | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 3- PET Scan 1 | 7.22 | NA — Data was not reported because only two participants were enrolled in this arm. | 4.80 | NA — Data was not reported because only two participants were enrolled in this arm. | 7.13 | NA — Data was not reported because only one participant was included in this arm.
  Participant 3- PET Scan 2 | 5.13 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.01 | NA — Data was not reported because only two participants were enrolled in this arm. | 7.46 | NA — Data was not reported because only one participant was included in this arm.
  Participant 3-PET Scan 3 | 4.53 | NA — Data was not reported because only two participants were enrolled in this arm. | 3.53 | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 4- PET Scan 1 | 7.37 | NA — Data was not reported because only two participants were enrolled in this arm. | 4.84 | NA — Data was not reported because only two participants were enrolled in this arm. | 7.48 | NA — Data was not reported because only one participant was included in this arm.
  Participant 4- PET Scan 2 | 2.72 | NA — Data was not reported because only two participants were enrolled in this arm. | 0.37 | NA — Data was not reported because only two participants were enrolled in this arm. | 4.35 | NA — Data was not reported because only one participant was included in this arm.
  Participant 4-PET Scan 3 | 11.13 | NA — Data was not reported because only two participants were enrolled in this arm. | 3.38 | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 1 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 3.69 | NA — Data was not reported because only two participants were enrolled in this arm. | 5.30 | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 2 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — PET scan 2 was not performed due to ligand synthesis failure. | NA — Data was not reported because only two participants were enrolled in this arm. | 6.38 | NA — Data was not reported because only one participant was included in this arm.
  Participant 5- PET Scan 3 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — PET scan 3 was not performed due to ligand synthesis failure. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data not reported since only PET Scan 1 and 2 were planned to be analyzed in Set B. | NA — Data was not reported because only one participant was included in this arm.
  Participant 6- PET Scan 1 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only five participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | 8.29 | NA — Data was not reported because only one participant was included in this arm.
  Participant 6- PET Scan 2 | NA — Data was not reported because only four participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data was not reported because only five participants were enrolled in this arm. | NA — Data was not reported because only two participants were enrolled in this arm. | NA — Data is not available because this participant withdrew the study after PET Scan 1. | NA — Data was not reported because only one participant was included in this arm.

3. Primary Outcome: D-amino Acid Oxidase (DAO) Occupancy Estimation in the Cerebellar GM
Description: DAO occupancy is calculated as percent difference between baseline and postdose [18F]PGM299 BPND for each participant.
Time Frame: as for outcome 1
Population: Due to variability in localization of [18F]PGM299 in both Cerebellar GM and Frontal Cortex GM, DAO occupancy estimation as a percent difference from baseline and post-TAK-831 dosing PET scans in Cerebellar GM based on VT values could not be made.
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg | Set A: [18F]PGM299 Baseline
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Set A: EC50- Plasma Concentration of TAK-831 That Corresponds to 50 Percent (%) DAO Brain Enzyme Occupancy in Cerebellum
Description: EC50 was obtained from global VT model. The affinity constant relating plasma concentration of TAK-831 to DAO occupancy (EC50) was estimated by fitting the PET and plasma concentration data (VT, Cp). It was calculated as VT= VsBase (EC50/EC50+Cp) + VND, where Vs Base was the group-level (global) volume of distribution of the specific binding in the target region (cerebellar GM) and VND was the volume of distribution of the non-displaceable component (non-specific bound and free radiotracer) of the target region.
Time Frame: Set A: Baseline, 2 and 26 hours post-TAK-831 dose
Population: The PET target occupancy set included all participants who received study drug (TAK-831) and had a technically adequate baseline PET scan and at least 1 technically adequate post-TAK-831 dose PET scan.
Measure: Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Groups:
- Set A: All Participants: Participants received TAK-831 100, 200, 250 or 500 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline, 2 hours and 26 hours post-TAK-831 dose.
Arm/Group | Set A: All Participants
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL) | 12.7 [2.3 to 23.1]

5. Secondary Outcome: Set A: Dose of TAK-831 That Corresponds to 50% DAO Brain Enzyme Occupancy in Cerebellum
Description: Dose of TAK-831 that corresponds to 50% DAO brain enzyme occupancy in cerebellum at the time of maximum observed plasma concentration (Tmax) of TAK-831 was estimated.
Time Frame: Set A: At 2 and 26 hours post-TAK-831 dose
Population: as for outcome 4
Measure: Number; unit: mg
Arm/Group | Set A: All Participants
Number analyzed (Participants) | 12
mg | 100

6. Secondary Outcome: Set B: Coefficient of Variation (CoV) of [18F]PGM299 Binding in Healthy Human Brain
Description: CoV was calculated as COV (P)(%) = 100 * mean/ standard deviation, where P was different participant scanned under baseline condition.
Time Frame: Set B: Baseline up to Day 10
Population: The analysis set included all participants in Set B who had completed technically evaluable test and re-test PET scans.
Measure: Number; unit: percentage of CoV
Arm/Group | Set B: [18F]PGM299
Number analyzed (Participants) | 5
percentage of CoV | 30.13

7. Secondary Outcome: Set A: Plasma Concentrations of TAK-831 During Each Post-TAK-831 Dosing PET Scan Periods
Time Frame: Set A: Days 1 and 2 At time 0 (at tracer injection), 60 minutes after tracer injection and 120 minutes after tracer injection for each post TAK-831 dosing PET scan period
Population: Pharmacokinetic(PK) set where data at specified time points post-tracer injection was available.PK set included all participants who received study drug(TAK-831)and had at least 1 measurable plasma concentration for TAK-831.Data was reported for Participant 1,2,3 and 4 of each of TAK-831 100,250mg and Participant 1 and 2 of TAK-831 200,500mg arms.
Measure: Mean (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 4 | 2
nanogram per milliliter (ng/mL)
  Day 1: pre-tracer dose | 211.250 [163.00 to 271.00] | 416.500 [201.00 to 632.00] | 273.750 [168.00 to 321.00] | 1404.500 [889.00 to 1920.00]
  Day 1: 60 minutes post-tracer dose | 83.375 [55.40 to 95.80] | 129.050 [78.10 to 180.00] | 122.725 [68.90 to 196.00] | 376.500 [254.00 to 499.00]
  Day 1: 120 minutes post-tracer dose | 42.500 [24.70 to 48.70] | 82.000 [64.00 to 100.00] | 89.925 [46.00 to 176.00] | 176.000 [130.00 to 222.00]
  Day 2: pre-tracer dose | 4.028 [2.74 to 7.21] | 7.360 [5.89 to 8.83] | 11.025 [8.17 to 14.20] | 23.400 [12.70 to 34.10]
  Day 2: 60 minutes post-tracer dose | 3.140 [1.62 to 5.74] | 5.205 [4.41 to 6.00] | 9.658 [6.60 to 13.80] | 28.455 [9.61 to 47.30]
  Day 2: 120 minutes post-tracer dose | 3.123 [1.26 to 5.89] | 5.380 [3.82 to 6.94] | 8.665 [5.70 to 14.60] | 33.975 [8.15 to 59.80]

8. Secondary Outcome: Set A: Percent Change From Baseline to Post-TAK-831 Dose in AUEC(0-24)Serine: Area Under the Effect-time Curve From Time 0 to 24 Hours Post-TAK-831 Dose for Dextro-serine (D-serine) and Levo-serine (L-serine)
Time Frame: Set A: Baseline, 24 hours post-TAK-831 dose
Population: The pharmacodynamic (PD) set for D- and L-serine included all participants in Set A who received study drug (TAK-831) and had at least 1 measurable D- and L-serine plasma measurement both at pre-dose and following TAK-831 dosing.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
percent change
  D-serine | 8.65 (7.209) | 21.90 (NA) — Standard deviation (SD) could not be estimated because only two participants were enrolled in this arm. | 18.08 (8.309) | 8.70 (NA) — SD could not be estimated because only two participants were enrolled in this arm.
  L-serine | 10.88 (5.905) | 2.00 (NA) — SD could not be estimated because only two participants were enrolled in this arm. | -2.46 (10.301) | 5.10 (NA) — SD could not be estimated because only two participants were enrolled in this arm.

9. Secondary Outcome: Set A: Percent Change From Baseline to Post-TAK-831 Dose in AUEC(0-24)Serine: Area Under the Effect-time Curve From Time 0 to 24 Hours Post-TAK-831 Dose for Ratio of D-serine to Total Serine
Time Frame: Set A: Baseline, 24 hours post-TAK-831 dose
Population: The PD set for D- and L-serine included all participants in Set A who received study drug (TAK-831) and had at least 1 measurable D- and L-serine plasma measurement both at pre-dose and following TAK-831 dosing.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
percent change | -1.18 (4.748) | 19.75 (NA) — SD could not be estimated because only two participants were enrolled in this arm. | 21.30 (6.958) | 6.25 (NA) — SD could not be estimated because only two participants were enrolled in this arm.

10. Secondary Outcome: Set A: Percent Change in Maximum Drug-induced Effect (Emax,Serine) on Change in Plasma Concentrations of D-serine and L-serine
Time Frame: Set A: Baseline, 24 hours post-TAK-831 dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
percent change
  D-serine | 9.58 (9.769) | 27.05 (NA) — SD could not be estimated because only two participants were enrolled in this arm. | 17.46 (9.122) | 40.30 (NA) — SD could not be estimated because only two participants were enrolled in this arm.
  L-serine | 17.40 (7.318) | 11.50 (NA) — SD could not be estimated because only two participants were enrolled in this arm. | -2.02 (12.917) | 16.10 (NA) — SD could not be estimated because only two participants were enrolled in this arm.

11. Secondary Outcome: Set A: Percent Change in Maximum Drug-induced Effect (Emax, D: Total Serine Ratio) on the Ratio of D-serine to Total Serine
Time Frame: Set A: Baseline, 24 hours post-TAK-831 dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
percent change | -1.40 (9.515) | 20.95 (NA) — SD could not be estimated because only two participants were enrolled in this arm. | 25.38 (12.604) | 20.45 (NA) — SD could not be estimated because only two participants were enrolled in this arm.

12. Secondary Outcome: Set A: Time to Reach the Maximum PD Effect (Time to Emax,Serine) for D-serine and L-serine
Time Frame: Set A: Day -1 At 1, 4 and 12 hours post check-in and Day 1 pre-dose and at multiple time points (up to 24 hours) post-TAK-831 dose
Population: The PD set for D- and L-serine included all participants in Set A who received study drug (TAK-831) and had at least 1 measurable D- and L-serine plasma measurement both at pre-dose and following TAK-831 dosing. PD set where data at specified time points were available.
Measure: Mean (Full Range); unit: hours
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
hours
  D-serine: Day -1: number analyzed (Participants) | 4 | 2 | 5 | 1
  D-serine: Day -1 | 4.955 [1.00 to 12.00] | 1.000 [1.00 to 1.00] | 3.320 [1.00 to 10.60] | 11.900 [11.90 to NA] — Maximum value could not be calculated, because only one participant in this arm.
  D-serine: Day 1 | 18.000 [12.00 to 20.00] | 18.000 [12.00 to 24.00] | 15.206 [4.03 to 20.00] | 25.100 [20.00 to 30.20]
  L-serine: Day -1: number analyzed (Participants) | 3 | 2 | 5 | 1
  L-serine: Day -1 | 4.267 [1.00 to 10.80] | 5.750 [1.00 to 10.50] | 6.086 [2.33 to 10.60] | 2.350 [2.35 to NA] — Maximum value could not be calculated, because only one participant in this arm.
  L-serine: Day 1: number analyzed (Participants) | 4 | 2 | 5 | 1
  L-serine: Day 1 | 13.993 [3.97 to 20.00] | 24.000 [24.00 to 24.00] | 12.026 [4.03 to 20.00] | 30.200 [30.20 to NA] — Maximum value could not be calculated, because only one participant in this arm.

13. Secondary Outcome: Set A: Time to Reach the Maximum PD Effect (Time to Emax,Serine) for Ratio of D-serine to Total Serine
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Full Range); unit: hours
Arm/Group | Set A: TAK-831 100 mg | Set A: TAK-831 200 mg | Set A: TAK-831 250 mg | Set A: TAK-831 500 mg
Number analyzed (Participants) | 4 | 2 | 5 | 2
hours
  Day -1: number analyzed (Participants) | 4 | 1 | 4 | 2
  Day -1 | 6.875 [1.00 to 12.00] | 1.000 [1.00 to NA] — Maximum value could not be calculated, because only one participant in this arm. | 1.875 [1.00 to 2.50] | 11.100 [10.30 to 11.90]
  Day 1 | 26.725 [23.60 to 29.90] | 25.000 [20.00 to 30.00] | 23.750 [8.05 to 30.40] | 30.100 [30.00 to 30.20]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to Day 15 in set A and up to Day 12 in set B.
Description: At each visit, investigator had to document any occurrence of adverse events and abnormal laboratory findings.Any event spontaneously reported by participant/observed by investigator was recorded,irrespective of relation to study treatment.
Groups:
- Set A: [18F]PGM299 Dose 1 to Prior TAK-831 100 mg Dose: [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline; and prior to TAK-831 100 mg, suspension, orally, once on Day 1.
- Set A: [18F]PGM299 Dose 1 to Prior TAK-831 200 mg Dose: [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline; and prior to TAK-831 200 mg, suspension, orally, once on Day 1.
- Set A: [18F]PGM299 Dose 1 to Prior TAK-831 250 mg Dose: [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline; and prior to TAK-831 250 mg, suspension, orally, once on Day 1.
- Set A: [18F]PGM299 Dose 1 to Prior TAK-831 500 mg Dose: [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at Baseline; and prior to TAK-831 500 mg, suspension, orally, once on Day 1.
- Set A: TAK-831 100 mg Dose to Prior [18F]PGM299 Dose 2: TAK-831 100 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at [18F]PGM299 Dose 2 (2 hours post-TAK-831 dose).
- Set A: TAK-831 200 mg Dose to Prior [18F]PGM299 Dose 2: TAK-831 200 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 18F]PGM299 Dose 2 (2 hours post-TAK-831 dose).
- Set A: TAK-831 250 mg Dose to Prior [18F]PGM299 Dose 2: TAK-831 250 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 18F]PGM299 Dose 2 (2 hours post-TAK-831 dose).
- Set A: TAK-831 500 mg Dose to Prior [18F]PGM299 Dose 2: TAK-831 500 mg, suspension, orally, once on Day 1 and up to 100 MBq of [18F]PGM299 with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 18F]PGM299 Dose 2 (2 hours post-TAK-831 dose).
- SetA:TAK-831 100mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15): [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 26 hours post-TAK-831 100 mg dose up to follow up on Day 15.
- SetA:TAK-831 200mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15): [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 26 hours post-TAK-831 200 mg dose up to follow up on Day 15.
- SetA:TAK-831 250mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15): [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 26 hours post-TAK-831 250 mg dose up to follow up on Day 15.
- SetA:TAK-831 500mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15): [18F]PGM299 up to 100 MBq with a maximal mass up to 12.5 mcg, injection, intravenously, prior to PET imaging at 26 hours post-TAK-831 500 mg dose up to follow up on Day 15.
Arm/Group | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 100 mg Dose | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 200 mg Dose | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 250 mg Dose | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 500 mg Dose | Set A: TAK-831 100 mg Dose to Prior [18F]PGM299 Dose 2 | Set A: TAK-831 200 mg Dose to Prior [18F]PGM299 Dose 2 | Set A: TAK-831 250 mg Dose to Prior [18F]PGM299 Dose 2 | Set A: TAK-831 500 mg Dose to Prior [18F]PGM299 Dose 2 | SetA:TAK-831 100mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) | SetA:TAK-831 200mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) | SetA:TAK-831 250mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) | SetA:TAK-831 500mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) | Set B: [18F]PGM299 | Set A: [18F]PGM299 Baseline
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/5 | 0/2 | 0/4 | 0/2 | 0/5 | 0/2 | 0/4 | 0/2 | 0/5 | 0/2 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 2/4 | 0/2 | 1/5 | 0/2 | 0/4 | 0/2 | 2/5 | 1/2 | 2/4 | 0/2 | 0/5 | 1/2 | 0/6 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 100 mg Dose (N=4) | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 200 mg Dose (N=2) | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 250 mg Dose (N=5) | Set A: [18F]PGM299 Dose 1 to Prior TAK-831 500 mg Dose (N=2) | Set A: TAK-831 100 mg Dose to Prior [18F]PGM299 Dose 2 (N=4) | Set A: TAK-831 200 mg Dose to Prior [18F]PGM299 Dose 2 (N=2) | Set A: TAK-831 250 mg Dose to Prior [18F]PGM299 Dose 2 (N=5) | Set A: TAK-831 500 mg Dose to Prior [18F]PGM299 Dose 2 (N=2) | SetA:TAK-831 100mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) (N=4) | SetA:TAK-831 200mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) (N=2) | SetA:TAK-831 250mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) (N=5) | SetA:TAK-831 500mg:[18F]PGM299 Dose 3 up to Follow-up (Day 15) (N=2) | Set B: [18F]PGM299 (N=6) | Set A: [18F]PGM299 Baseline (N=1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.